CLINICAL TRIAL: NCT01857921
Title: Combination Effects of High-dose Statin and Trimetazidine on Patients With Aspirin Mono Antiplatelet Therapy 12-months After Coronary Artery Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2010-0511
Record Dates: First submitted 2013-05-15; First posted 2013-05-20 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2018-12

CONDITIONS: Coronary Artery
MeSH Terms: interventions — Pravastatin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pravastatin group (Active Comparator)
  Interventions: Drug: Pravastatin 20mg/day for 12 months after randomization
- Combination of Atorvastatin and trimetazidine group (Experimental)
  Interventions: Drug: Atorvastatin 40 mg and trimetazidine MR 70 mg/day for 12 months after randomization

INTERVENTIONS:
Drug: Pravastatin 20mg/day for 12 months after randomization — Patients with mono antiplatelet therapy with aspirin who had had received CABG previously fulfilling all enrollment criteria will be randomly assigned to the type of two groups. Randomization of statin therapy will be done 1:1 to one of two different groups on the web-based program:
  1. Test group:
     * Atorvastatin 40 mg and trimetazidine MR 70 mg daily for 12 months after randomization
  2. Control group:
     * Pravastatin 20mg daily for 12 months after randomization
  Arms: Pravastatin group
Drug: Atorvastatin 40 mg and trimetazidine MR 70 mg/day for 12 months after randomization — Patients with mono antiplatelet therapy with aspirin who had had received CABG previously fulfilling all enrollment criteria will be randomly assigned to the type of two groups. Randomization of statin therapy will be done 1:1 to one of two different groups on the web-based program:
  1. Test group:
     * Atorvastatin 40 mg and trimetazidine MR 70 mg daily for 12 months after randomization
  2. Control group:
     * Pravastatin 20mg daily for 12 months after randomization
  Arms: Combination of Atorvastatin and trimetazidine group

SUMMARY:
Trimetazidine is a metabolic agent without any negative inotropic or vasodilatory properties. In addition, previous reports showed that trimetazidine was effective in reducing intracoronary platelet aggregation and preventing platelet thrombogenesis. Therefore, for the evaluation of these combination effects of statin and trimetazidine on patients with aspirin monotherapy who had previously received CABG and were free of the major adverse cardiac events such as death, MI, TLR, or TVR for 12 months, the investigators hypothesize that atorvastatin 40mg/day would be more effective in the prevention of the further late adverse cardiac and cerebrovascular events than other statin. To test this hypothesis, the investigators will perform a multi-center, randomized, prospective trial aimed at demonstrating the superiority of combination of high dose atorvastatin therapy and trimetazidine to pravastatin in patients with aspirin monotherapy 12 months after CABG surgery in real world practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had previously received CABG 12 months ago
* Patients who were free of death, MI or repeat revascularization within first 12 months after CABG
* Patients with mono antiplatelet therapy with aspirin alone
* Age of 20 years or older
* Patients with signed informed consent

Exclusion Criteria:

* History of DES or BMS implantation within 12 months
* Patients who required the continuing dual antiplatelet therapy or additional other types of antithrombotics or antiplatelets such as cilostazol or ticlopidine, etc besides aspirin after DES implantation
* Patients who could not be prescribed aspirin or statins due to contraindication or severe side effects
* Pregnant women or women with potential childbearing
* Life expectancy ≤ 2 year

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2010-12; Primary Completion 2018-04-08 (Actual); Study Completion 2018-04-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of the composite of death from any cause | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea